CLINICAL TRIAL: NCT00606528
Title: FGL2/Fibroleukin and Hepatitis C Virus Infection: A Predictor of Response to Antiviral Therapy
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0841-T
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Antiviral therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Plasma Liver tissue from biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: patients with chronic Hepatitis C Virus infection who have not previously received antiviral therapy
  Interventions: Other: No intervention
- Group B: Healthy volunteers willing to donate blood on 2 separate occasions

INTERVENTIONS:
Other: No intervention — None. This is an observational study.
  Groups: Group A

SUMMARY:
The main objective of this study is to assess whether a recently-developed bioassay for the protein FGL2 can be used to predict the progression and/or response to treatment of Hepatitis C Virus disease in patients with chronic HCV infection. The hypothesis is that increased levels of FGL2 and increased numbers of T regulatory cells are associated with a failure to respond to treatment.

DETAILED DESCRIPTION:
The current therapy for chronic Hepatitis C Virus infection leads to a sustained viral response in only 50% of treated patients. Evidence suggests that a poor response to treatment may be the result of a dysfunction of immunoregulatory mediators including T regulatory cells (Tregs) which secrete FGL2. The aim of this study is to test whether serum FGL2 levels can serve as a biomarker for clinical progress and treatment response in patients undergoing anti-viral therapy for chronic HCV infection.

This study will measure the blood Treg and FGL2 levels of patients with chronic Hepatitis C as they undergo antiviral therapy and will compare those levels to their pre-treatment and post-treatment levels. Treg and FGL2 expression levels will also be measured in patients' liver biopsy tissue when available.

Additionally, this study will examine the main form(s)of Fc Receptor expressed in these patients. The Fc receptor is the hypothesized binding partner of FGL2, and the form expressed in a given patient may determine the downstream effects of FGL2's binding. These data along with clinical, biochemical and virological data will be used to determine whether there is a correlation between FGL2 levels and disease outcome and/or treatment response.

The study will also recruit a group of normal healthy volunteers to give blood samples on two occasions so that the baseline range of FGL2 levels in healthy individuals can be established for comparison.

ELIGIBILITY:
HCV patient population

Inclusion Criteria:

* able to give written consent
* 18-70 yrs of age, both genders
* willing to use adequate contraception
* diagnosis of chronic HCV infection (of any genotype) based on 2 positive serology tests
* availability of pre- and post-treatment viral load data
* naive to antiviral treatment
* availability of pre-treatment liver biopsy

Exclusion Criteria:

* less than 18 yrs, greater than 70 yrs of age
* pregnancy
* HBV, HDV, or HIV co-infection
* any history of active alcohol or drug abuse

Volunteer Population (Control)

Inclusion Criteria:

* able and willing to provide written informed consent
* willing to provide a brief review of medical history
* 18-70 yrs of age, of either gender

Exclusion Criteria:

* less than 18, greater than 70 yrs of age
* any history of liver, renal, lung, hematological or coronary artery disease
* any history of active alcohol or drug abuse
* any previous diagnosis of HBV, HCV, HDV or HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic HCV treatment-naive patients who are willing to begin antiviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
correlation between blood FGL2 levels and response to antiviral therapy | 6 months after the end of treatment

SECONDARY OUTCOMES:
correlation between FGL2 levels and Treg percentage in blood and liver cells | all time points

CONTACTS AND LOCATIONS:
Overall Officials: Gary Levy, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Shalev I, Liu H, Koscik C, Bartczak A, Javadi M, Wong KM, Maknojia A, He W, Liu MF, Diao J, Winter E, Manuel J, McCarthy D, Cattral M, Gommerman J, Clark DA, Phillips MJ, Gorczynski RR, Zhang L, Downey G, Grant D, Cybulsky MI, Levy G. Targeted deletion of fgl2 leads to impaired regulatory T cell activity and development of autoimmune glomerulonephritis. J Immunol. 2008 Jan 1;180(1):249-60. doi: 10.4049/jimmunol.180.1.249. PMID 18097026
- [Background] Liu H, Zhang L, Cybulsky M, Gorczynski R, Crookshank J, Manuel J, Grant D, Levy G. Identification of the receptor for FGL2 and implications for susceptibility to mouse hepatitis virus (MHV-3)-induced fulminant hepatitis. Adv Exp Med Biol. 2006;581:421-5. doi: 10.1007/978-0-387-33012-9_76. No abstract available. PMID 17037572
- [Background] Chan CW, Kay LS, Khadaroo RG, Chan MW, Lakatoo S, Young KJ, Zhang L, Gorczynski RM, Cattral M, Rotstein O, Levy GA. Soluble fibrinogen-like protein 2/fibroleukin exhibits immunosuppressive properties: suppressing T cell proliferation and inhibiting maturation of bone marrow-derived dendritic cells. J Immunol. 2003 Apr 15;170(8):4036-44. doi: 10.4049/jimmunol.170.8.4036. PMID 12682232